CLINICAL TRIAL: NCT02255565
Title: Quillivant XR in Children With Attention Deficit/Hyperactivity Disorder (ADHD) and Autism Spectrum Disorder (ASD): A Pilot Study
Brief Title: Dose Response Effects of Quillivant XR in Children With ADHD and Autism: A Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Mark Stein, Director of ADHD/Related Disorders Program, Seattle Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WI185890
Record Dates: First submitted 2014-09-24; First posted 2014-10-02 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: ADHD; Autism
Keywords: Quillivant
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autistic Disorder | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Very Low Dose Quillivant XR (Experimental): Patients in this treatment arm are given Quillivant XR (a liquid medication) to treat ADHD at a very low dose level for 6 weeks.
  Interventions: Drug: Very Low Dose Quillivant XR
- Low Dose Quillivant XR (Experimental): Patients in this treatment arm are given Quillivant XR (a liquid medication) to treat ADHD at a low dose level for 6 weeks.
  Interventions: Drug: Low Dose Quillivant XR
- Moderate dose Quillivant XR (Experimental): Patients in this treatment arm are given Quillivant XR (a liquid medication) to treat ADHD at a moderate dose level for 6 weeks.
  Interventions: Drug: Moderate Dose Quillivant XR

INTERVENTIONS:
Drug: Very Low Dose Quillivant XR — Oral suspension dose once a day increasing to a 10mg dose
  Other Names: Methylphenidate HCl
  Arms: Very Low Dose Quillivant XR
Drug: Low Dose Quillivant XR — Oral suspension dose once a day increasing to a 20mg dose
  Other Names: Methylphenidate HCl
  Arms: Low Dose Quillivant XR
Drug: Moderate Dose Quillivant XR — Oral suspension dose once a day increasing to a 40mg dose
  Other Names: Methylphenidate HCl
  Arms: Moderate dose Quillivant XR

SUMMARY:
The purpose of this study is to determine whether Quillivant XR is effective in the treatment of ADHD in children with Autism Spectrum Disorder (ASD).

DETAILED DESCRIPTION:
To evaluate the safety and tolerability of low to moderate dose effects of Quillivant XR (liquid methylphenidate) and to observe changes in ADHD symptoms and functional outcomes in children with ASD and ADHD. The investigators propose to investigate the low to moderate dose range of methylphenidate compared with a very low dose with a gradual dose escalation schedule because children with ASD have been found to be more sensitive to the adverse effects of methylphenidate (especially in medium to high doses) than children without ASD.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of Autistic disorder or Asperger's disorder by DSM-IV or Autism Spectrum Disorder by DSM-V.
* A DSM-V diagnosis of ADHD based upon the K-SADS-P.
* Clinical Global Impressions - Severity for ADHD (CGI-S-ADHD) rating > 4.
* Findings on physical exam, labs and ECG are judged to be normal for age with pulse and blood pressure within 95% of age and gender mean.
* Informed consent by a parent or legal guardian, and assent for children with developmental age 7 years or older.
* At least one parent fluent in English

Exclusion Criteria:

* History of Seizure disorder (Febrile seizures are non-exclusionary).
* History of Intellectual Disability (IQ< 70)
* Treatment with MAO Inhibitor (or within 14 days following discontinuation of MAO Inhibitor).
* Other psychotropic medication other than stable dose of Selective Serotonin Reuptake Inhibitors, which is permitted)
* Known to be hypersensitive to methylphenidate, or other components of Quillivant XR
* Cardiac or other medical contraindications for stimulant trial (e.g., family history of heart attack at age younger than 40 years, personal history of heart disease, history of fainting while exercising, structural cardiac abnormalities, cardiomyopathy, serious cardiac arrhythmias, coronary artery disease, or other serious cardiac problems. If any doubt, children will be referred to a cardiologist for a cardiac clearance.
* Raynaud's disease
* Pregnancy or Breast-feeding.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2014-09; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stein, PhD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

REFERENCES:
- [Background] Gadow KD, DeVincent CJ, Pomeroy J. ADHD symptom subtypes in children with pervasive developmental disorder. J Autism Dev Disord. 2006 Feb;36(2):271-83. doi: 10.1007/s10803-005-0060-3. PMID 16477513
- [Background] Lee DO, Ousley OY. Attention-deficit hyperactivity disorder symptoms in a clinic sample of children and adolescents with pervasive developmental disorders. J Child Adolesc Psychopharmacol. 2006 Dec;16(6):737-46. doi: 10.1089/cap.2006.16.737. PMID 17201617
- [Background] Rao, P. A. and R. J. Landa (2013).
- [Background] Research Units on Pediatric Psychopharmacology Autism Network. Randomized, controlled, crossover trial of methylphenidate in pervasive developmental disorders with hyperactivity. Arch Gen Psychiatry. 2005 Nov;62(11):1266-74. doi: 10.1001/archpsyc.62.11.1266. PMID 16275814
- [Background] Stein, M.A. et al.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were recruited from the investigators' practices, clinic referrals, and letter mailings. Participants were enrolled between September 2014 and September 2016.
Pre-assignment Details: Of the 36 participants enrolled, 27 were randomized to receive treatment. 3 participants withdrew, 2 due to time commitment issues and 1 due to stress over screening. 6 participants were deemed ineligible for the study due to no Autism Spectrum Disorder (ASD) diagnosis based on screening assessments.
Groups:
- Very Low Dose Quillivant XR: Patients in this treatment arm are given Quillivant XR (a liquid medication) to treat ADHD at a very low dose level for 6 weeks.
  Very Low Dose Quillivant XR: Oral suspension dose once a day starting at 5mg and increasing to a 10mg dose
- Low Dose Quillivant XR: Patients in this treatment arm are given Quillivant XR (a liquid medication) to treat ADHD at a low dose level for 6 weeks.
  Low Dose Quillivant XR: Oral suspension dose once a day starting at 5mg and increasing to a 20mg dose
- Moderate Dose Quillivant XR: Patients in this treatment arm are given Quillivant XR (a liquid medication) to treat ADHD at a moderate dose level for 6 weeks.
  Moderate Dose Quillivant XR: Oral suspension dose once a day starting at 5mg and increasing to a 40mg dose
Period: Overall Study
Arm/Group | Very Low Dose Quillivant XR | Low Dose Quillivant XR | Moderate Dose Quillivant XR
Started | 9 | 9 | 9
Completed | 9 | 8 | 9
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Of the 36 participants enrolled, 27 were randomized to receive treatment. 3 participants withdrew, 2 due to time commitment issues and 1 due to stress over screening. 6 participants were deemed ineligible for the study due to no Autism Spectrum Disorder (ASD) diagnosis based on screening assessments.
Groups:
- Total: Total of all reporting groups
Arm/Group | Very Low Dose Quillivant XR | Low Dose Quillivant XR | Moderate Dose Quillivant XR | Total
Number analyzed (Participants) | 9 | 9 | 9 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 9 | 9 | 27
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.33 (2.92) | 8.00 (2.96) | 10.22 (3.03) | 9.19 (3.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2
  Male | 8 | 9 | 8 | 25
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 9 | 26

OUTCOME MEASURES:

1. Primary Outcome: ADHD Rating Scale - IV
Description: Measures the severity of Total ADHD symptoms, Inattention and Hyperactivity/Impulsive symptoms. The Inattention and Hyperactivity/Impulsive symptoms can range from 0 to 27 each, with a higher score reflecting more severe ADHD symptoms. The total score is calculated by summing the inattention and Hyperactivity/Impulsive subscales. The total score can range from 0 to 54 with a higher score reflecting more severe ADHD symptoms.
Time Frame: once a week for 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Very Low Dose Quillivant XR - Week 1; Very Low Dose Quillivant XR - Week 2; Very Low Dose Quillivant XR - Week 3; Very Low Dose Quillivant XR - Week 4; Very Low Dose Quillivant XR - Week 5; Very Low Dose Quillivant XR - Week 6: Patients in this treatment arm are given Quillivant XR (a liquid medication) to treat ADHD at a very low dose level for 6 weeks. The dose titration was based on the physician's discretion and parent-reported Adverse Events (AE's).
  Very Low Dose Quillivant XR: Oral suspension dose once a day starting at 5mg and increasing to a 10mg dose
- Low Dose Quillivant XR - Week 1; Low Dose Quillivant XR - Week 2; Low Dose Quillivant XR - Week 3; Low Dose Quillivant XR - Week 4; Low Dose Quillivant XR - Week 5; Low Dose Quillivant XR - Week 6: Patients in this treatment arm are given Quillivant XR (a liquid medication) to treat ADHD at a low dose level for 6 weeks.The dose titration was based on the physician's discretion and parent-reported Adverse Events (AE's).
  Low Dose Quillivant XR: Oral suspension dose once a day starting at 5mg and increasing to a 20mg dose
- Moderate Dose Quillivant XR - Week 1; Moderate Dose Quillivant XR - Week 2; Moderate Dose Quillivant XR - Week 3; Moderate Dose Quillivant XR - Week 4; Moderate Dose Quillivant XR - Week 5; Moderate Dose Quillivant XR - Week 6: Patients in this treatment arm are given Quillivant XR (a liquid medication) to treat ADHD at a moderate dose level for 6 weeks. The dose titration was based on the physician's discretion and parent-reported Adverse Events (AE's).
  Moderate Dose Quillivant XR: Oral suspension dose once a day starting at 5mg and increasing to a 40mg dose
Arm/Group | Very Low Dose Quillivant XR - Week 1 | Very Low Dose Quillivant XR - Week 2 | Very Low Dose Quillivant XR - Week 3 | Very Low Dose Quillivant XR - Week 4 | Very Low Dose Quillivant XR - Week 5 | Very Low Dose Quillivant XR - Week 6 | Low Dose Quillivant XR - Week 1 | Low Dose Quillivant XR - Week 2 | Low Dose Quillivant XR - Week 3 | Low Dose Quillivant XR - Week 4 | Low Dose Quillivant XR - Week 5 | Low Dose Quillivant XR - Week 6 | Moderate Dose Quillivant XR - Week 1 | Moderate Dose Quillivant XR - Week 2 | Moderate Dose Quillivant XR - Week 3 | Moderate Dose Quillivant XR - Week 4 | Moderate Dose Quillivant XR - Week 5 | Moderate Dose Quillivant XR - Week 6
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 8 | 8 | 9 | 9 | 9 | 9 | 9 | 9 | 9
units on a scale
  Inattention Subscale Score | 17.89 (3.95) | 16.78 (4.18) | 16.67 (2.74) | 14.33 (6.26) | 14.56 (5.53) | 12.89 (5.01) | 16.33 (6.89) | 14.00 (5.83) | 12.00 (5.22) | 8.38 (5.90) | 9.50 (4.57) | 9.56 (6.17) | 18.11 (4.43) | 14.67 (5.15) | 13.67 (6.98) | 13.56 (5.10) | 13.00 (5.55) | 11.78 (5.43)
  Hyperactivity Subscale Score | 12.44 (7.91) | 10.56 (8.16) | 11.56 (6.25) | 12.33 (5.70) | 9.22 (7.55) | 8.78 (5.67) | 15.33 (8.23) | 14.33 (7.38) | 10.22 (5.24) | 6.88 (4.42) | 9.38 (4.75) | 6.56 (4.28) | 12.78 (3.87) | 11.33 (2.78) | 11.78 (6.26) | 9.67 (5.87) | 9.22 (5.83) | 7.33 (2.87)
  Total Score | 30.33 (9.27) | 27.33 (11.14) | 28.22 (7.24) | 26.67 (10.20) | 23.78 (11.51) | 21.67 (7.78) | 31.67 (14.67) | 28.33 (12.41) | 22.22 (9.90) | 15.25 (9.77) | 18.88 (9.06) | 16.11 (8.99) | 30.89 (6.17) | 26.00 (5.87) | 25.44 (12.70) | 23.22 (10.02) | 22.22 (10.03) | 19.11 (7.44)

2. Secondary Outcome: Clinical Global Impressions-ADHD - Severity
Description: The CGI-S scale summarizes the clinician's impression of the participant's symptom severity and ranges from 1-7 with 1 representing normal (not at all ill) and 7 representing extremely ill.
Time Frame: once a week for 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Low Dose Quillivant XR - Week 1; Low Dose Quillivant XR - Week 2; Low Dose Quillivant XR - Week 3; Low Dose Quillivant XR - Week 4; Low Dose Quillivant XR - Week 5; Low Dose Quillivant XR - Week 6: Patients in this treatment arm are given Quillivant XR (a liquid medication) to treat ADHD at a low dose level for 6 weeks. The dose titration was based on the physician's discretion and parent-reported Adverse Events (AE's).
  Low Dose Quillivant XR: Oral suspension dose once a day starting at 5mg and increasing to a 20mg dose
- Moderate Dose Quillivant XR - Week 1; Moderate Dose Quillivant XR - Week 2; Moderate Dose Quillivant XR - Week 3; Moderate Dose Quillivant XR - Week 4; Moderate Dose Quillivant XR - Week 5; Moderate Dose Quillivant XR - Week 6: Patients in this treatment arm are given Quillivant XR (a liquid medication) to treat ADHD at a low dose level for 6 weeks. The dose titration was based on the physician's discretion and parent-reported Adverse Events (AE's).
  Low Dose Quillivant XR: Oral suspension dose once a day starting at 5mg and increasing to a 40mg dose
Arm/Group | Very Low Dose Quillivant XR - Week 1 | Very Low Dose Quillivant XR - Week 2 | Very Low Dose Quillivant XR - Week 3 | Very Low Dose Quillivant XR - Week 4 | Very Low Dose Quillivant XR - Week 5 | Very Low Dose Quillivant XR - Week 6 | Low Dose Quillivant XR - Week 1 | Low Dose Quillivant XR - Week 2 | Low Dose Quillivant XR - Week 3 | Low Dose Quillivant XR - Week 4 | Low Dose Quillivant XR - Week 5 | Low Dose Quillivant XR - Week 6 | Moderate Dose Quillivant XR - Week 1 | Moderate Dose Quillivant XR - Week 2 | Moderate Dose Quillivant XR - Week 3 | Moderate Dose Quillivant XR - Week 4 | Moderate Dose Quillivant XR - Week 5 | Moderate Dose Quillivant XR - Week 6
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 8 | 8 | 9 | 9 | 9 | 9 | 9 | 9 | 9
units on a scale | 4.78 (0.44) | 4.33 (0.87) | 4.44 (0.88) | 4.33 (0.87) | 4.11 (1.05) | 4.00 (0.87) | 4.33 (1.12) | 4.00 (1.22) | 3.67 (1.00) | 2.75 (1.16) | 2.88 (1.25) | 2.78 (1.30) | 4.89 (0.33) | 4.56 (0.53) | 4.11 (0.60) | 4.00 (0.71) | 3.56 (0.88) | 3.44 (1.24)

3. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I)
Description: The CGI-I scale summarizes the clinician's impression of the participant's symptom improvement and ranges from 1-7 with 1 representing very much improved and 7 representing very much worse.
Time Frame: once a week for 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Very Low Dose Quillivant XR - Week 1; Very Low Dose Quillivant XR - Week 2; Very Low Dose Quillivant XR - Week 3; Very Low Dose Quillivant XR - Week 4; Very Low Dose Quillivant XR - Week 5; Very Low Dose Quillivant XR - Week 6: Patients in this treatment arm are given Quillivant XR (a liquid medication) to treat ADHD at a low dose level for 6 weeks. The dose titration was based on the physician's discretion and parent-reported Adverse Events (AE's).
  Low Dose Quillivant XR: Oral suspension dose once a day starting at 5mg and increasing to a 10mg dose
Arm/Group | Very Low Dose Quillivant XR - Week 1 | Very Low Dose Quillivant XR - Week 2 | Very Low Dose Quillivant XR - Week 3 | Very Low Dose Quillivant XR - Week 4 | Very Low Dose Quillivant XR - Week 5 | Very Low Dose Quillivant XR - Week 6 | Low Dose Quillivant XR - Week 1 | Low Dose Quillivant XR - Week 2 | Low Dose Quillivant XR - Week 3 | Low Dose Quillivant XR - Week 4 | Low Dose Quillivant XR - Week 5 | Low Dose Quillivant XR - Week 6 | Moderate Dose Quillivant XR - Week 1 | Moderate Dose Quillivant XR - Week 2 | Moderate Dose Quillivant XR - Week 3 | Moderate Dose Quillivant XR - Week 4 | Moderate Dose Quillivant XR - Week 5 | Moderate Dose Quillivant XR - Week 6
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 9 | 8 | 8 | 9 | 9 | 9 | 9 | 9 | 9 | 9
units on a scale | 3.89 (0.60) | 3.56 (0.88) | 3.44 (0.53) | 3.22 (0.83) | 3.00 (1.00) | 2.89 (0.78) | 3.78 (1.30) | 3.00 (0.87) | 2.22 (0.83) | 1.63 (0.74) | 2.13 (0.99) | 2.00 (0.87) | 3.33 (0.50) | 3.11 (0.60) | 2.67 (1.12) | 2.89 (0.60) | 2.56 (1.01) | 2.22 (0.83)

ADVERSE EVENTS:
Time Frame: 6 weeks. Adverse events were collected from participants while they were in the study, this time frame was 6 weeks.
Description: At each weekly visit, children and their parents met with the investigators and research staff. Parents completed the Response Impressions Side Effects Checklist - Kids (RISK Checklist), a 38-item scale that is rated on a 10-point (0-9) scale ranging from absent to serious.
Arm/Group | Very Low Dose Quillivant XR | Low Dose Quillivant XR | Moderate Dose Quillivant XR
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 8/9 | 8/9 | 9/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Very Low Dose Quillivant XR (N=9) | Low Dose Quillivant XR (N=9) | Moderate Dose Quillivant XR (N=9)
Difficulty Falling Asleep (General disorders) | 5 (17) | 6 (10) | 6 (17)
Waking at Night (General disorders) | 2 (2) | 2 (5) | 1 (1) — Difficulty remaining asleep throughout the night
Waking up Early (General disorders) | 3 (9) | 5 (16) | 2 (5) — Premature awakening in the morning, is too alert to resume sleeping after waking
Nightmares (General disorders) | 1 (1) | 0 (0) | 1 (1) — Distressing dreams
Flat Affect / No Emotion (Psychiatric disorders) | 2 (3) | 0 (0) | 2 (2) — Complete (or nearly complete) absence of emotional expression.
Rebound at end of day (Psychiatric disorders) | 4 (16) | 4 (19) | 5 (15) — An intensification of ADHD symptoms at the end of the day
Aggression (Psychiatric disorders) | 6 (16) | 2 (5) | 4 (7) — Behaving in an actively hostile manner
Talks less (General disorders) | 2 (3) | 1 (1) | 2 (2) — Child talks less than is normal for him/her.
Uninterested (General disorders) | 2 (7) | 1 (1) | 4 (5) — Child appears not to be interested in things or people around him/her
Decreased Appetite (General disorders) | 3 (9) | 6 (13) | 4 (13) — Reduction in the intensity or frequency of hunger; a reduced desire to eat
Irritable (General disorders) | 7 (22) | 4 (6) | 4 (11) — Easily irritated or annoyed
Hostility (General disorders) | 6 (18) | 3 (5) | 5 (7) — Showing antagonism and opposition towards people and/or circumstances
Stomachaches (General disorders) | 2 (2) | 2 (2) | 0 (0) — Persistent pain localized in the stomach area
Headaches (General disorders) | 2 (2) | 0 (0) | 0 (0) — Persistent physical pain in the child's head
Drowsiness (General disorders) | 1 (1) | 2 (3) | 3 (3) — An irresistible urge to fall asleep at inappropriate times
Sad/Unhappy (General disorders) | 1 (1) | 1 (1) | 0 (0) — Child appears inappropriately sad (moods is not congruent with setting or circumstance)
Prone to Crying (General disorders) | 4 (12) | 3 (8) | 1 (2) — Cries easily or often
Anxious/worries (General disorders) | 3 (11) | 3 (8) | 2 (2) — Apprehension, fear, concern, or dread
Bites Fingernails (General disorders) | 2 (7) | 1 (1) | 1 (1) — Child bites fingernails or cuticles
Picking (General disorders) | 1 (1) | 1 (1) | 3 (9) — Child picks at skin, cuticles, fingernails, etc.
Euphoric/Happy (General disorders) | 3 (4) | 3 (9) | 5 (9) — Child appears inappropriately happy (mood is not congruent with setting or circumstance)
Nausea (General disorders) | 1 (1) | 2 (2) | 0 (0) — The urge to vomit; child feels like he/she might vomit
Tics (Psychiatric disorders) | 2 (8) | 2 (3) | 3 (4) — Child makes repetitive, uncontrollable movements or sounds
Jittery or nervous (General disorders) | 2 (6) | 2 (4) | 1 (1) — An edgy, tense state; is easily agitated or anxious
Mood Swings/Lability (General disorders) | 5 (17) | 3 (5) | 3 (5) — Unpredictable or easily changeable moods; unstable moods or emotions
Fatigue (General disorders) | 1 (1) | 2 (2) | 1 (3) — A reduction of strength or energy
Constipation (Gastrointestinal disorders) | 2 (7) | 3 (9) | 0 (0) — Infrequent bowel movements
Stares A Lot (General disorders) | 0 (0) | 2 (2) | 3 (3) — Child frequently has a fixed look with his/her wide open, looks into space
Abdominal pain (General disorders) | 0 (0) | 1 (1) | 0 (0) — Persistent pain localized in the abdomen
Rash (General disorders) | 0 (0) | 1 (1) | 3 (9) — Skin becomes reddened, itchy, and/or raised (not due to an insect bite)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Throwing up
Cold Hands and Feet (General disorders) | 0 (0) | 0 (0) | 1 (1) — Hands and feet are cold to the touch

LIMITATIONS AND CAVEATS:
No placebo was available for comparison to Quillivant XR. Small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No